CLINICAL TRIAL: NCT00886795
Title: A Phase I/II Open-label Study to Evaluate The Safety and Efficacy of Abatacept in Subjects With Chronic Urticaria Who Have Had an Inadequate Response to Anti-histamine Therapy.
Brief Title: Safety and Efficacy of Abatacept in Subjects With Chronic Urticaria Who Have Had an Inadequate Response to Anti-histamine Therapy
Acronym: TAHOE
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Principal Investigator, Clifton O Bingham, M.D., Johns Hopkins University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Tahoe-001
Record Dates: First submitted 2009-04-22; First posted 2009-04-23 (Estimated); Results first posted 2016-01-25 (Estimated); Last update posted 2016-01-25 (Estimated); Status verified 2015-12

CONDITIONS: Urticaria
Keywords: hives; rash; pruritis
MeSH Terms: conditions — Urticaria; Exanthema; Pruritus | interventions — Abatacept

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Abatacept (Experimental): 4 doses of abatacept administered intravenously at baseline, 2 weeks, 4 weeks, and 8 weeks.
  Interventions: Drug: abatacept (Orencia ®)

INTERVENTIONS:
Drug: abatacept (Orencia ®) — 4 doses of abatacept administered intravenously at baseline, 2 weeks, 4 week, and 8 weeks.
  Other Names: orencia

SUMMARY:
This study is being done to find out if a drug called Abatacept (Orencia ®) is safe and effective in treating people with chronic urticaria (persistent hives).

ELIGIBILITY:
Inclusion Criteria:

* Chronic active urticaria defined as symptoms > 50% of days or 3 days/week for more than 12 weeks
* Chronic therapy with stable doses of antihistamines for at least 4 weeks (patients may be taking more than one antihistamine or be taking combinations of antihistamines and leukotriene receptor antagonists) AND failure to respond to at least maximally approved dosages of 2 different antihistamine therapies
* One of the following 3 conditions:

  * Previous or ongoing requirement for corticosteroids for symptom control OR
  * Prior steroid treatment with steroid discontinuation due to unacceptable morbidity
  * Previous or current use (without symptom control or with unacceptable morbidity: e.g., hypertension from cyclosporine, hemolysis from dapsone) of immunomodulatory treatment for urticaria (e.g., hydroxychloroquine, methotrexate, sulfasalazine, dapsone, cyclosporine, intravenous immunoglobulin (IVIg), mycophenolate, azathioprine, etc)
* High baseline score for pruritis (at least 2 on a 3 point scale)
* No underlying etiology clearly defined for urticaria
* Patients should exhibit evidence of underlying autoimmunity of at least one of the following:

  * elevated erythrocyte sedimentation rate (ESR), C-Reactive Protein (CRP), anti-nuclear antibody (ANA)
  * extractable nuclear antigens
  * Thyroid antibodies
  * other autoantibodies (e.g., intrinsic factor, parietal cell, ovarian), *elevated complement levels
  * clinical characteristics suggestive of systemic autoimmune disease but without satisfying criteria for another diagnosis (e.g., arthralgias, myalgias, arthritis, low grade fever, significant fatigue associated with outbreaks)
  * family history of autoimmune disease including thyroid autoimmunity
  * a biopsy showing perivascular lymphocytic or mixed cellular infiltrate without vasculitis
* Concomitant use of hydroxychloroquine, methotrexate, or sulfasalazine will be permitted if dose stable for at least 8 weeks
* Concomitant use of steroids (≤ 15 mg/d Prednisone or equivalent) will be permitted if stable for 4 weeks and patient agrees to continue dose for the first 90 days
* Negative pregnancy test (for women of child-bearing age)
* Men and women of reproductive potential must agree to use an acceptable birth control during treatment and for 3 months after treatment
* No planned elective surgical procedures for at least 6 months from day#1

Exclusion Criteria:

* Current use of other immunosuppressive medications (cyclosporine, tacrolimus, sirolimus, IVIg, cyclophosphamide, mycophenolate mofetil, azathioprine). Any such medication will be discontinued for at least 4 weeks before study drug start.
* Concomitant treatment with corticosteroids (≤ 15 mg/d), hydroxychloroquine, methotrexate, and sulfasalazine will be permitted if doses are stable at least 8 weeks
* Treatment with an investigational agent within 4 weeks of screening or 5 half-lives of the investigational drug (whichever is longer)
* Receipt of a live vaccine within 4 weeks of randomization
* Prior treatment with Abatacept (Orencia®)
* Previous treatment with Rituximab (MabThera®/Rituxan®), unless 6 months after administration AND B cell reconstitution has occurred into normal range
* History of severe allergic or anaphylactic reactions to monoclonal antibodies or Fc fusion proteins
* History of significant laryngeal edema, tongue swelling, or airway compromise in the setting of urticarial/angioedema episode (isolated perioral, lip, and periorbital edema will not be exclusionary)
* Known history of Human Immunodeficiency Virus (HIV), Hepatitis B and/or Hepatitis C
* purified protein derivative (PPD) testing as part of screening that is positive*
* HIV, Hepatitis B surface antigen or Core Antibody positive, or anti Hepatitis C Antibody positive detected with screening
* History of recurrent significant infection, active bacterial, viral, fungal, mycobacterial, or other infection excluding fungal infections of nail beds, or major infection requiring hospitalization or treatment with IV antibiotics within 4 weeks of screening or oral antibiotics within 2 wks of screening
* Known immunodeficiency, hypogammaglobulinemia, etc.
* Systemic lupus erythematosus (meeting American College of Rheumatology (ACR)) criteria; patients with autoantibodies such as ANA will NOT be excluded)
* Lack of peripheral venous access
* Drug, alcohol, or chemical abuse within 6 months
* Pregnancy or lactation and all women must be willing to practice contraception through the study duration and for 3 months after discontinuing abatacept treatment.

  * Sexually active women of childbearing potential must use an effective method of birth control during the course of the study, in a manner such that risk of failure is minimized.
  * Prior to study enrollment, women of childbearing potential (WOCBP) will be advised of the importance of avoiding pregnancy during trial participation and the potential risk factors for an unintentional pregnancy.
  * In addition, men enrolled on this study will be informed of the risks to any sexual partner of childbearing potential and counseled to practice an effective method of birth control.
  * All WOCBP must have a negative urine pregnancy test within 7 days prior to first receiving the investigational product.
  * If the pregnancy test is positive, the subject will be excluded from the study.
  * In addition, all WOCBP will be instructed to contact the Investigator immediately if they suspect they might be pregnant (e.g., missed or late menstrual period) at any time during study participation and the Investigator will notify Bristol Myers Squibb (BMS) within 24 hours of becoming aware of a confirmed pregnancy in a subject participating in the study.
  * Women must agree to practice adequate birth control for a minimum of 3 months post-treatment.
* Concomitant malignancies or previous malignancies within five years, with exception of adequately treated basal or squamous cell carcinoma of the skin or carcinoma in situ of cervix
* Atopic dermatitis, psoriasis, or autoimmune bullous skin disease (pemphigus, pemphigoid, etc)
* Significant cardiovascular disease (angina, arrhythmia, known coronary artery disease, cerebrovascular accident (CVA), transient ischemic attack (TIA), uncontrolled hypertension > 150/90)
* Significant pulmonary disease (asthma or chronic obstructive pulmonary disease (COPD) requiring current use of corticosteroids, history ever of severe asthma or status asthmatics)
* Any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates an investigational drug or that may affect interpretation of the results or render patient at high risk from treatment complications
* Plans or need to receive live viral vaccination over course of the study (e.g., Flu-Mist)
* Inability to comply with study and follow-up procedures

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2009-05; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clifton O. Bingham, M.D., Principal Investigator — Associate Professor of Medicine
Locations (1):
- Johns Hopkins Arthritis Center, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Abatacept: 4 doses of abatacept administered intravenously at baseline, 2 weeks, 4 weeks, and 8 weeks.
  abatacept (Orencia ®): 4 infusions of abatacept administered intravenously at baseline, 2 weeks, 4 week, and 8 weeks. The dose of abatacept received by each participant was based on weight. Participants received either 500mg, 750mg , or 1000mg of abatacept based on weights of >60 kg, 60-100kg, or 100 kg respectively.
Period: Overall Study
Arm/Group | Abatacept
Started | 4
Completed | 3
Not Completed | 1
Not completed — Lack of Efficacy | 1

BASELINE CHARACTERISTICS:
Groups:
- Abatacept: 4 doses of abatacept administered intravenously at baseline, 2 weeks, 4 weeks, and 8 weeks.
  abatacept (Orencia ®): 4 doses of abatacept administered intravenously at baseline, 2 weeks, 4 week, and 8 weeks.The dose of abatacept received by each participant was based on weight. Participants received either 500mg, 750mg , or 1000mg of abatacept based on weights of >60 kg, 60-100kg, or 100 kg respectively.
Arm/Group | Abatacept
Number analyzed (Participants) | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 43 (7.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: Participants were monitored for adverse events (AEs) at each visit. Cumulative AEs were tracked including specific AE, severity, and relationship on source documentation. Special attention was given to infusion-related events and hypersensitivity reactions. Assessment of Complete Blood Count (CBC) and Metabolic profile were also tracked.
Time Frame: baseline, 3 month and 6 months
Population: Participants who received all four doses.
Measure: Number; unit: participants
Arm/Group | Abatacept
Number analyzed (Participants) | 4
participants | 3

2. Secondary Outcome: Number of Participants With Clinically Detectable Improvement
Description: Evaluations will occur at each visit after the first infusion. At 3 months, response will be recorded and patients with improvement will be eligible to move into the steroid and/or antihistamine tapering portion of the study. Improvement was determined by a reduction in the number of hives.
Time Frame: at each visit and at 3 months
Measure: Number; unit: participants
Arm/Group | Abatacept
Number analyzed (Participants) | 4
participants | 4

ADVERSE EVENTS:
Time Frame: 3 years
Description: Adverse events were collected by patient report at each study visit in response to open ended questioning.
Arm/Group | Abatacept
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 3/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Abatacept (N=4)
Headache (Nervous system disorders) | 2 (3)
Common Cold (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Influenza (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Diastasis (Musculoskeletal and connective tissue disorders) | 1 (1)
Ear Infection (Infections and infestations) | 1 (1)
Hypoesthesia (Nervous system disorders) | 1 (1)
Right Shoulder Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Rhinorrhea (General disorders) | 1 (1)
Sinus Infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Tinea Pedis (Skin and subcutaneous tissue disorders) | 1 (1)
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Open Label study. Small number of patients. Outcome measures for urticaria not standardized.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less